CLINICAL TRIAL: NCT02453165
Title: Randomized Clinical Trial About Vaginal Cuff Dehiscence Following Total Laparoscopic Hysterectomy: Laparoscopic vs. Transvaginal Cuff Suturing
Brief Title: Vaginal Cuff Dehiscence Following Total Laparoscopic Hysterectomy: Laparoscopic vs. Transvaginal Cuff Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Stefano Uccella, Medical Doctor, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 440
Record Dates: First submitted 2015-02-03; First posted 2015-05-25 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Surgical Wound Dehiscence
Keywords: vaginal dehiscence
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRANSVAGINAL SUTURE (Experimental): INTERVENTION: Transvaginal suturE of the vaginal vault at the end of a total laparoscopic hysterectomy using vaginal valves and needleholders.
  Interventions: Procedure: TRANSVAGINAL SUTURE
- LAPAROSCOPIC SUTURE (Active Comparator): INTERVENTION: Laparoscopic suturE of the vaginal vault at the end of a total laparoscopic hysterectomy using with laparoscopic needleholders.
  Interventions: Procedure: LAPAROSCOPIC SUTURE

INTERVENTIONS:
Procedure: TRANSVAGINAL SUTURE — The closure of the vaginal cuff will be performed transvaginally using a 0-poly-g-lactin braided and coated medium-term reabsorbable suture with vaginal valves and needleholders
  Arms: TRANSVAGINAL SUTURE
Procedure: LAPAROSCOPIC SUTURE — The closure of the vaginal cuff will be performed laparoscopically using a 0-poly-g-lactin braided and coated medium-term reabsorbable suture with laparoscopic needleholders
  Arms: LAPAROSCOPIC SUTURE

SUMMARY:
Post-hysterectomy vaginal cuff dehiscence is a rare but threatening complication.

The investigators will compare transvaginal versus laparoscopic closure of the vaginal vault at the end of a total laparoscopic hysterectomy, in order which of these two modalities of suturing is associated with a lower risk of dehiscence.

DETAILED DESCRIPTION:
A post-hysterectomy vaginal cuff dehiscence is defined as a partial or total separation of the margins of the vaginal cuff closure, following hysterectomy.

The recognition of the complication is made on a clinical basis. The investigators will compare the percentage of dehiscence among women who had transvaginal vs. laparoscopic suture of the vault.

The investigators will also compare the two modalities in terms of:

* duration of the vaginal closure
* risk of bleeding from the vaginal cuff
* risk of post-operative pelvic infection
* risk of re-operation
* dyspareunia
* total vaginal length
* vaginal cuff prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total laparoscopic hysterectomy with or without salpingo-oophorectomy

Exclusion Criteria:

* Patients with gynecological malignancy (uterine and/or adnexal)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1408 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
VAGINAL DEHISCENCE | 3 months postoperatively
  Vaginal dehiscence defined as any partial or complete separation of the vaginal vault, sutured at the end of a total laparoscopic hysterectomy.
  This complication is diagnosed clinically, during a gynecologic visit. Every dehiscence (whether partial or total) will be considered as an outcome event and we will measure the presence/absence of dehiscence as a percentage of the total procedures.

SECONDARY OUTCOMES:
VAGINAL CUFF COMPLICATIONS | 3 months postoperatively
  * Vaginal bleeding
  * Need for Vaginal re-suture
  * Vaginal vault prolapse
  * Dyspareunia
  * Post-operative pelvic infection
operative time | During Operation
  Time spent in suturing the vaginal cuff transvaginally vs. laparoscopically

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Uccella, MD, PhD, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- Department of Obstetrics and Gynecology Universita' Dell'Insubria, Varese, Italy

REFERENCES:
- [Result] Ceccaroni M, Berretta R, Malzoni M, Scioscia M, Roviglione G, Spagnolo E, Rolla M, Farina A, Malzoni C, De Iaco P, Minelli L, Bovicelli L. Vaginal cuff dehiscence after hysterectomy: a multicenter retrospective study. Eur J Obstet Gynecol Reprod Biol. 2011 Oct;158(2):308-13. doi: 10.1016/j.ejogrb.2011.05.013. Epub 2011 Jul 1. PMID 21723030
- [Result] Hur HC, Donnellan N, Mansuria S, Barber RE, Guido R, Lee T. Vaginal cuff dehiscence after different modes of hysterectomy. Obstet Gynecol. 2011 Oct;118(4):794-801. doi: 10.1097/AOG.0b013e31822f1c92. PMID 21934442
- [Result] Uccella S, Ghezzi F, Mariani A, Cromi A, Bogani G, Serati M, Bolis P. Vaginal cuff closure after minimally invasive hysterectomy: our experience and systematic review of the literature. Am J Obstet Gynecol. 2011 Aug;205(2):119.e1-12. doi: 10.1016/j.ajog.2011.03.024. Epub 2011 Mar 22. PMID 21620360
- [Result] Uccella S, Ceccaroni M, Cromi A, Malzoni M, Berretta R, De Iaco P, Roviglione G, Bogani G, Minelli L, Ghezzi F. Vaginal cuff dehiscence in a series of 12,398 hysterectomies: effect of different types of colpotomy and vaginal closure. Obstet Gynecol. 2012 Sep;120(3):516-23. doi: 10.1097/AOG.0b013e318264f848. PMID 22914459
- [Result] Kim MJ, Kim S, Bae HS, Lee JK, Lee NW, Song JY. Evaluation of risk factors of vaginal cuff dehiscence after hysterectomy. Obstet Gynecol Sci. 2014 Mar;57(2):136-43. doi: 10.5468/ogs.2014.57.2.136. Epub 2014 Mar 15. PMID 24678487
- [Result] Nieboer TE, Johnson N, Lethaby A, Tavender E, Curr E, Garry R, van Voorst S, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD003677. doi: 10.1002/14651858.CD003677.pub4. PMID 19588344
- [Derived] Uccella S, Capozzi VA, Ricco' M, Perrone E, Zanello M, Ferrari S, Zorzato PC, Seracchioli R, Cromi A, Serati M, Ergasti R, Fanfani F, Berretta R, Malzoni M, Cianci S, Vizza E, Guido M, Legge F, Ciravolo G, Gueli Alletti S, Ghezzi F, Candiani M, Scambia G. Sexual Function following Laparoscopic versus Transvaginal Closure of the Vaginal Vault after Laparoscopic Hysterectomy: Secondary Analysis of a Randomized Trial by the Italian Society of Gynecological Endoscopy Using a Validated Questionnaire. J Minim Invasive Gynecol. 2020 Jan;27(1):186-194. doi: 10.1016/j.jmig.2019.03.018. Epub 2019 Apr 3. PMID 30951920